CLINICAL TRIAL: NCT04192604
Title: Development and Validation of the Work-related MusculoSkeletal Disorders Risk Assessment Questionnaire
Brief Title: Work-related MusculoSkeletal Disorders Questionnaire
Acronym: WMSD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: WMSDsQ
Record Dates: First submitted 2019-11-21; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Musculoskeletal Diseases; Work-Related Condition
Keywords: Work-related musculoskeletal pain; pain management; prevention; screening
MeSH Terms: conditions — Musculoskeletal Diseases; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: WMSDsQ — Work-related MusculoSkeletal Disorders Questionnaire

SUMMARY:
Development and validation of a multi-factor and self-perceived risk assessment questionnaire, specifically referred to WMSDs-related pain and risk factors

DETAILED DESCRIPTION:
The World Health Organization (WHO) has defined a WMSD as one musculoskeletal disorder (MSD) that results from a number of factors, and where the work environment and the performance of the work contribute significantly, but in varying magnitude, to the causation of the disease. The term MSD denotes health problems of the musculoskeletal system, i.e. muscles, tendons, the skeleton, cartilage, the vascular system, ligaments and nerves; ranging from light and transitory disorders to disabling injuries and permanent disability, with the loss of employment. WMSDs are in general not caused by one specific, but by multiple risk factors. These include physical (e.g. manual handling of loads, working in awkward postures, repetitive work and working at high speed, exposure to vibrations) as well as psychosocial (work stress, pain believes, sleep disturbances) factors. Consequently, a holistic preventive approach is currently needed. In order to tackle WMSDs, three different levels of prevention can be used to categorise these strategies: i) primary prevention includes the risk assessment process and technical/ergonomic, organisational and person-oriented interventions; ii) secondary prevention involves the identification and health monitoring of workers at risk; and iii) tertiary prevention comprises return-to-work actions.

The answer to the WMSDs problems in companies is holistic prevention, taking into account multifactorial risks for every individual, in order to propose a tailored educational program to every worker need

The study aims to develop and validate a multi-factor and self-perceived risk assessment questionnaire, specifically referred to WMSDs-related pain and risk factors

Gathering information and collecting data on the target population and WMSDs related risk factors:

* Basic characteristics of the target populations (e.g. age, sex, work conditions etc.)
* Potential work-related risk factors (e.g. repetitive motion, static posture, etc.)
* Which of WMSDs affect more the target populations (e.g. back pain, neck pain, upper limb pain, etc.)
* Potential effects of these and related domains (quality of life, pain, number of days of absence from work etc.)

ELIGIBILITY:
Inclusion Criteria:

* Understanding of the Italian language
* Worker of the IRCCS Istituto Ortopedico Galeazzi

Exclusion Criteria:

- Previous surgery for musculoskeletal disorders

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The sample size was set at 115 subjects. This number was established on the basis of available data deriving from surveys previously carried out in the same type of population.
  The test-retest will be submitted to 20 subjects. The sample will be selected randomly from a numerical generator at intervals between 1 and n (with n = highest registration number of the center workers) among the workers of the IRCCS Istituto Ortopedico Galeazzi. Furthermore, to obtain a homogeneous distribution, the sample will be evaluated according to the type of work and according to it will be stratified into 3 categories: health workers, administrative workers, other workers. The inclusion of the subjects in each category will be interrupted when they reach 40% of the total sample. In this way, the maximum possible inhomogeneity of the sample will be 40%-40%-20%.
Sampling Method: Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2020-01-15 (Estimated); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Development and validation | November 2019 - August 2020 (9 months)
  Development and validation of a multi-factor and self-perceived risk assessment questionnaire, specifically referred to WMSDs-related pain and risk factors

SECONDARY OUTCOMES:
Risk Factors | November 2019 - August 2020 (9 months)
  Estimation of potential work-related risk factors of WMSDs.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Langella F, Vanni D, Hogh M, Palsson TS, Christensen SWM, Bellosta-Lopez P, Villafane JH, Jensen PS, Silva PB, Herrero P, Barletta P, Domenech-Garcia V, Berjano P; Prevent for Work Study Group. Development of the Prevent for Work Questionnaire (P4Wq) for the assessment of musculoskeletal risk factors in the workplace: part 2-pilot study for questionnaire development and validation. BMJ Open. 2021 Dec 24;11(12):e053988. doi: 10.1136/bmjopen-2021-053988. PMID 34952882